CLINICAL TRIAL: NCT06189001
Title: The Role of Oxytocin-receptor Signalling in Physiological Regulation of Eating Behaviour in Individuals with Obesity
Acronym: FOxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-23059585
Record Dates: First submitted 2023-12-05; First posted 2024-01-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-05

CONDITIONS: Adiposity
Keywords: oxytocin; appetite regulation; gastrointestinal motility; energy expenditure
MeSH Terms: conditions — Obesity | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Intravenous oxytocin 0.2 IU/minute for 300 minutes Approx. 500 ml
  Interventions: Drug: Oxytocin
- Placebo (Other): intravenous saline (0.9% NaCl) infusion for 300 minutes Approx. 500 ml
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Drug: Oxytocin — Intravenous oxytocin 0.2 IU/min during experimental days
  Arms: Oxytocin
Other: Placebo (saline) — Intravenous saline during experimental days
  Arms: Placebo

SUMMARY:
The present study evaluates appetite, glucose metabolism, gastrointestinal motility and energy expenditure in men and women with obesity (BMI 30-40 kg/m2) under oxytocin exposure compared to placebo.

DETAILED DESCRIPTION:
In a randomised, double-blind, placebo-controlled, crossover fashion, 24 participants will complete two experimental days (A and B) including a mixed meal test and an ad libitum meal test. The procedures during the two experimental days are similar except for intravenous infusion of oxytocin on experimental day A and placebo (saline) on experimental day B, respectively. On experimental days, oxytocin or placebo infusion will be started at timepoint -60 minutes. At timepoint 0 minutes, participants will ingest a liquid mixed meal. After 190 minutes, participants are served an ad libitum meal followed by ad libitum snacks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI between 30 and 40 kg/m2 (both included)
* Percentage body fat (BF%) ≥25 for men and ≥32 for women (assessed by bioelectrical impedance analysis)
* Informed oral and written consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALT) >2 times normal values
* History of hepatobiliary and/or gastrointestinal disorder(s)
* Kidney disease (serum creatinine above normal range and/or urine albumin-creatinine ratio (uACR) >30 mg/g confirmed by two measures)
* Previous gastric or intestinal resection, cholecystectomy and/or any major intra-abdominal surgery (including bariatric surgery)
* Previous pancreatic disease and/or neoplasia
* Regular tobacco smoking and/or use of other nicotine products
* Glycated haemoglobin (HbA1c) ≥48 and/or type 1 diabetes or type 2 diabetes requiring medical treatment
* Pituitary gland disorders
* Initiation of special diets, lifestyle changes and/or weight loss >5% of total body weight within three months prior to or during study period
* Pregnancy or breastfeeding
* Long QTc on electrocardiogram (ECG) at screening (≥0.45 seconds for men and ≥0.46 seconds for women)
* Any physical or psychological condition or ongoing medication the investigator group suspect would interfere with trial participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake | Timepoint 190-220 minutes
  Amount consumed (kcal)

SECONDARY OUTCOMES:
Ad libitum food intake | Timepoint 190-220 minutes
  Amount consumed (kcal/kg)
Sensations of hunger | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of satiety | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of fullness | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of prospective food intake | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of nausea | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of thirst | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Sensations of comfort | Timepoint -100 to 160 minutes
  Visual analogue score (VAS) (0-100 mm) (bsAUC)
Composite appetite score | Timepoint -100 to 160
  Calculated from VAS of hunger, fullness and prospective food intake (bsAUC)
Plasma concentrations of glucose | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of glucose | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of glucose | Timepoint -95 to 180 minutes
  Peak value
Serum concentrations of insulin | Timepoint -95 to 180 minutes
  Baseline
Serum concentrations of insulin | Timepoint -95 to 180 minutes
  bsAUC
Serum concentrations of C-peptide | Timepoint -95 to 180 minutes
  Baseline
Serum concentrations of C-peptide | Timepoint -95 to 180 minutes
  bsAUC
Beta cell function (C-peptide/glucose-ratio) | Timepoint -95 to 180 minutes
  Baseline
Beta cell function (C-peptide/glucose-ratio) | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of cholecystokinin | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of cholecystokinin | Timepoint -95 to 180 minutes
  bsAUC
Energy expenditure (indirect calorimetry) | Timepoint -90 to 150 minutes
  Resting energy expenditure (REE)
Energy expenditure (indirect calorimetry) | Timepoint -90 to 150 minutes
  Respiration exchange rate (RER)
Snacking (ad libitum snack test) | Timepoint 225-235 minutes
  Amount consumed (kcal)
Gallbladder volume (ml) | Timepoint -120 to 180 minutes
  Baseline
Gallbladder volume (ml) | Timepoint -120 to 180 minutes
  AUC
Gallbladder ejection fraction (%) | Timepoint -120 to 180 minutes
  GBEF%
Gallbladder volume (ml) | Timepoint -120 to 180 minutes
  Nadir
Gallbladder volume | Timepoint -120 to 180 minutes
  Time to nadir (min)
Plasma concentrations of glucagon | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of glucagon | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of GLP-1 | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of GLP-1 | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of GIP | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of GIP | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of peptide YY | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of peptide YY | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of leptin | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of leptin | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of ghrelin | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of ghrelin | Timepoint -95 to 180 minutes
  bsAUC
Plasma concentrations of secretin | Timepoint -95 to 180 minutes
  Baseline
Plasma concentrations of secretin | Timepoint -95 to 180 minutes
  bsAUC
Gastric emptying (paracetamol absorption method) | Timepoint -95 to 180 minutes
  Baseline
Gastric emptying (paracetamol absorption method) | Timepoint -95 to 180 minutes
  bsAUC
Circulating levels of total amino acids | Timepoint -95 to 180 minutes
  Baseline
Circulating levels of total amino acids | Timepoint -95 to 180 minutes
  bsAUC
Lipid profile | Timepoint -95 to 180 minutes
  Baseline
Lipid profile | Timepoint -95 to 180 minutes
  bsAUC
Circulating levels of CTx | Timepoint -95 to 180 minutes
  Baseline
Circulating levels of CTx | Timepoint -95 to 180 minutes
  bsAUC
Circulating levels of P1NP | Timepoint -95 to 180 minutes
  Baseline
Circulating levels of P1NP | Timepoint -95 to 180 minutes
  bsAUC
Circulating levels of PTH | Timepoint -95 to 180 minutes
  Baseline
Circulating levels of PTH | Timepoint -95 to 180 minutes
  bsAUC
Circulating levels of calcium | Timepoint -95 to 180 minutes
  Baseline
Circulating levels of calcium | Timepoint -95 to 180 minutes
  bsAUC
Desire for specific foods | Timepoint -100 to 160 minutes
  VAS (0-100 mm). Baseline
Desire for specific foods | Timepoint -100 to 160 minutes
  VAS (0-100 mm). bsAUC
Duration of ad libitum meal | Timepoint 190-220 minutes
  Minutes
Water intake during ad libitum meal | Timepoint 190-220 minutes
  ml
Blood pressure | Timepoint -75 to 185 minutes and timpoint 240 minutes
  Baseline
Blood pressure | Timepoint -75 to 185 minutes and timpoint 240 minutes
  bsAUC
Heart rate | Timepoint -75 to 185 minutes and timpoint 240 minutes
  Baseline
Heart rate | Timepoint -75 to 185 minutes and timpoint 240 minutes
  bsAUC
Plasma concentrations of creatinine | Timepoint -95 and 235 minutes
  Baseline
Plasma concentrations of creatinine | Timepoint -95 and 235 minutes
  End-infusion
Plasma concentrations of potassium | Timepoint -95 and 235 minutes
  Baseline
Plasma concentrations of potassium | Timepoint -95 and 235 minutes
  bsAUC
Plasma concentrations of sodium | Timepoint -95 and 235 minutes
  Baseline
Plasma concentrations of sodium | Timepoint -95 and 235 minutes
  End-infusion
Happiness (Oxford Happiness Questionnaire (translated to Danish)) | Timepoint -65 and 160 minutes
  Points on scale from 29-174
Circulating levels of high-sensitive C-reactive protein (hsCRP) | Timepoint -95 and 235 minutes
  Baseline
Circulating levels of C-reactive protein (hsCRP) | Timepoint -95 and 235 minutes
  End-infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolisk Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No